CLINICAL TRIAL: NCT06483399
Title: Influence of Nutritional Risk Indexes and Inflammatory Indicators on Postoperative Complications and Prognosis of Epithelial Ovarian Cancer and Construction of Prediction Models
Brief Title: Research on Nutritional Risk Indexes and Inflammatory Indicators in Postoperative Complications and Prognosis of Epithelial Ovarian Cancer Patients
Status: Completed | Type: Observational
Sponsor: Qinglei Gao (Other)
Responsible Party: Sponsor-Investigator, Qinglei Gao, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 2024-TJ-NIOC
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low [index] group: The patients were grouped according to the cut-off value of each index, and the patients whose index value was lower than the cut-off value were classified as the Low [index] group.
- High [index] group: The patients were grouped according to the cut-off value of each index, and the patients whose index value was higher than the cut-off value were classified as the High [index] group.

SUMMARY:
The goal of this observational study is to explore the influence and predictive significance of nutritional risk indicators and inflammatory indicators on postoperative complications and prognosis of patients with epithelial ovarian cancer (EOC). The main question it aims to answer is:

Can preoperative nutritional risk and inflammatory indexes predict postoperative complications? Do preoperative nutritional risk and inflammatory indexes better predict the prognosis of patients with epithelial ovarian cancer? Which index is the best predictor of postoperative complications or prognosis for patients?

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed primary epithelial ovarian, peritoneal, and fallopian tube cancers.
2. patients received comprehensive staged surgery or debulking surgery.
3. available data of laboratory examination within 7 days before the surgery.

Exclusion Criteria:

1. borderline ovarian tumor.
2. receipt of neoadjuvant chemotherapy.
3. presence of other conditions influencing laboratory data, like hepatitis, kidney disease, autoimmune diseases, infectious diseases, blood disease, etc.
4. concurrent cancer in other organs.
5. absence of surgery or biopsy only.
6. multiple staged surgeries.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with epithelial ovarian cancer between January 2012 and February 2023 were recruited from seven tertiary medical centers in the China Real World Gynecological Oncology Platform (NUWA).
Sampling Method: Probability Sample
Enrollment: 1108 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Postoperative Complications | Within 30 days after surgery
  Surgical complications within 30 days after comprehensive staging or cytoreductive surgery recorded according to the Clavien-Dindo grading system
Progression-free survival | From the date the patient diagnosed with primary ovarian, fallopian tube, or peritoneal cancer to the date of disease progression or death or last follow-up, whichever occurred first, assessed up to 100 months.
  Interval between first diagnosis and first recurrence, death, or last follow-up
Overall survival | From the date the patient diagnosed with primary ovarian, fallopian tube, or peritoneal cancer to the date of death or last follow-up, whichever occurred first, assessed up to 100 months.
  Interval between first diagnosis and death, or last follow-up

REFERENCES:
- [Derived] Liu X, Li M, Zhao Y, Jiao X, Yu Y, Li R, Zeng S, Chi J, Ma G, Huo Y, Peng Z, Liu J, Zhou Q, Zou D, Wang L, Li Q, Wang J, Yao S, Chen Y, Ma D, Hu T, Gao Q. The impact of preoperative immunonutritional status on postoperative complications in ovarian cancer. J Ovarian Res. 2025 Apr 29;18(1):88. doi: 10.1186/s13048-025-01624-3. PMID 40301987